CLINICAL TRIAL: NCT02256969
Title: Prospective, Randomized Clinical Trial of Meibomian Gland Probing Versus Sham Procedure for Refractory Meibomian Gland Dysfunction
Brief Title: Intraductal Meibomian Gland Probing Trial
Acronym: MGP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph B. Ciolino, MD (Other)
Responsible Party: Sponsor-Investigator, Joseph B. Ciolino, MD, Assistant Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-059H
Record Dates: First submitted 2014-08-13; First posted 2014-10-06 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — sulfanizolone; Sulfacetamide; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Meibomian Gland Probing plus lubricant (Other): Meibomian Gland Probing: Stainless steel probes were used to probe all the meibomian glands of upper lids of both eyes at the slit lamp. All patients were probed with a 1-mm probe followed by a 2-mm probe for all glands.
  Lubricant: GenTeal PM Night-Time Ointment (Alcon), a sterile ophthalmic lubricant that is commonly used to relieve symptoms in patients with dry eye disease, was applied topically to both eyes for 4 weeks with the following regimen: twice daily for 2 weeks and then once daily for 2 weeks.
  Interventions: Drug: GenTeal PM Night-Time; Procedure: Meibomian Gland Probing
- Sham Meibomian Gland Probing plus lubricant (Other): Sham Meibomian Gland Probing: The patient's the lid margin was touched with the probes without actual probing occurring.
  Lubricant: GenTeal PM Night-Time Ointment, ophthalmic lubricant used to relieve symptoms in patients with dry eye disease, was applied topically to both eyes for 4 weeks: twice daily for 2 weeks and then once daily for 2 weeks.
  Interventions: Drug: GenTeal PM Night-Time; Procedure: Sham Meibomian Gland Probing
- Meibomian Gland Probing plus Blephamide (Active Comparator): Meibomian Gland Probing: Stainless steel probes were used to probe all the meibomian glands of upper lids of both eyes at the slit lamp. All patients were probed with a 1-mm probe followed by a 2-mm probe for all glands.
  Blephamide: is a combination of an antibiotic and an anti-inflammatory agent commonly used to treat various ocular conditions. Blephamide was applied topically to both eyes for 4 weeks with a regimen of: twice daily for 2 weeks and then once daily for 2 weeks.
  Interventions: Drug: Blephamide; Procedure: Meibomian Gland Probing

INTERVENTIONS:
Drug: Blephamide
  Other Names: sulfacetamide sodium 10%/prednisolone acetate 0.2%, Allergan, Inc.
  Arms: Meibomian Gland Probing plus Blephamide
Drug: GenTeal PM Night-Time
  Other Names: GenTeal PM Night-Time Ophthalmic Ointment Alcon
  Arms: Meibomian Gland Probing plus lubricant; Sham Meibomian Gland Probing plus lubricant
Procedure: Meibomian Gland Probing — For anesthesia, topical 3.5% lidocaine hydrochloride jelly (Akron) was applied directly with sterile cotton-tipped applicator to the lid margin for 3 times every 10 minutes before the procedure. If necessary, 2% lidocaine was injected into the lid margin during the procedure to provide additional comfort. After obtaining adequate anesthesia, the solid stainless steel probes (Maskin® Meibomian Gland Intraductal Probes, Rhein Medical Inc.) were used to probe all the meibomian glands of upper lids of both eyes at the slit lamp. All patients were initially be probed with a 1-mm probe followed by a 2-mm probe for all glands.
  Arms: Meibomian Gland Probing plus Blephamide; Meibomian Gland Probing plus lubricant
Procedure: Sham Meibomian Gland Probing — For anesthesia, topical 3.5% lidocaine hydrochloride jelly (Akron) was applied directly with sterile cotton-tipped applicator to the lid margin for 3 times every 10 minutes before the procedure. If necessary, 2% lidocaine was injected into the lid margin during the procedure to provide additional comfort. The patient's lid margin was touched with the probes without actual probing of the meibomian gland orifices.
  Arms: Sham Meibomian Gland Probing plus lubricant

SUMMARY:
In this research study, the investigators are looking at the effects of Meibomian Gland Probing (MGP) versus a sham (fake) procedure in patients with refractory MGD who have already tried traditional management with no success in resolving their clinical signs (as seen by their ophthalmologist) or their symptoms.

The investigators are also evaluating the effects of using two (2) post-procedural medication treatments: Blephamide or GenTeal PM Night-Time to determine if treatment after the MGP procedure has an effect on its outcome.

DETAILED DESCRIPTION:
Dry eye disease is one of the most common conditions seen in ophthalmic practice and is associated with significant patient distress. Meibomian gland dysfunction (MGD) is among the most prevalent causes of dry eye disease. This condition, which is often due to obstruction of the meibomian gland orifices, may result in significant ocular irritation. Traditionally, management of MGD includes warm compress, lid hygiene, and anti-inflammatory medications. This randomized clinical trial is designed to evaluate the effects of meibomian gland probing versus sham procedure in cases with refractory MGD that do not respond to traditional treatments. Moreover, the effects of postoperative regimen will also be investigated using two different regimens. In addition to symptoms, the changes will also be evaluated in terms of clinical signs as well as in vivo confocal microscopy (IVCM) which allows study at the cellular level.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89 years
* Willing and able to provide written informed consent
* Willing and able to comply with study assessments for the full duration of the study
* Diagnosis of meibomian gland dysfunction (MGD)
* Symptoms of MGD such as foreign body sensation, burning, stinging, light sensitivity for at least 3 months
* Persistent symptoms despite at least 3 months of medical management including lid hygiene, warm compress, and use of topical and systemic therapy, or contraindication to systemic therapy
* Presence of lid tenderness on the upper lids in both eyes
* Tear break-up time (TBUT) of <10 seconds
* In good stable overall health

Exclusion Criteria:

* Active allergies to steroids, sulfacetamide, GenTeal PM Night-Time ointment, or lidocaine
* Intraocular surgery or ocular laser surgery within 1 month before enrollment
* History of ocular infection within 1 month before enrollment.
* History of increased intraocular pressure after using topical steroids (steroid responsive)
* Any condition (including language barrier) that precludes subject's ability to comply with study requirements including completion of study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Ciolino, M. D., Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kheirkhah A, Kobashi H, Girgis J, Jamali A, Ciolino JB, Hamrah P. A randomized, sham-controlled trial of intraductal meibomian gland probing with or without topical antibiotic/steroid for obstructive meibomian gland dysfunction. Ocul Surf. 2020 Oct;18(4):852-856. doi: 10.1016/j.jtos.2020.08.008. Epub 2020 Aug 31. PMID 32882429

RESULTS

PARTICIPANT FLOW:
Groups:
- Meibomian Gland Probing Plus Lubricant: Meibomian Gland Probing: Stainless steel probes were used to probe all the meibomian glands of upper lids of both eyes at the slit lamp.
  Lubricant: GenTeal PM Night-Time Ointment, an ophthalmic lubricant that is used to relieve symptoms in patients with dry eye disease; was applied topically to both eyes for 4 weeks: twice daily for 2 weeks and then once daily for 2 weeks.
- Meibomian Gland Probing Plus Blephamide: Meibomian Gland Probing: Stainless steel probes were used to probe the meibomian glands of upper lids of both eyes. All patients were probed with a 1-mm probe followed by a 2-mm probe for all glands.
  Blephamide: is a combination of an antibiotic and an anti-inflammatory agent commonly used to treat various ocular conditions. Blephamide was applied topically to both eyes for 4 weeks with a regimen of: twice daily for 2 weeks and then once daily for 2 weeks.
Period: Overall Study
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide
Started | 15 | 15 | 15
Completed | 13 | 14 | 14
Not Completed | 2 | 1 | 1
Not completed — Screenfailed or withdrew | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide | Total
Number analyzed (Participants) | 13 | 14 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13.7) | 63.9 (13.8) | 59.8 (17.4) | 61.1 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 3 | 4 | 5 | 12
Ocular Surface Disease Index (OSDI) [Mean (Standard Deviation); unit: units on a scale] — The overall ODSI score is calculated by adding all of the values from the 12 questions, multiplying that value by 25, and dividing the resulting value by the number of questions answered. This results in an overall scale that ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms.
  units on a scale | 45.3 (23.8) | 49.1 (27.1) | 49.1 (19.9) | 47.9 (23.3)
Symptom Assessment in Dry Eye (SANDE) [Mean (Standard Deviation); unit: units on a scale] — A two-item survey used to assess the frequency and severity of dry eye disease. The SANDE score is calculated by taking the square root of the product of the frequency of symptoms score and the severity of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
  units on a scale | 68.7 (15.4) | 61.8 (22.5) | 72.1 (14.1) | 67.5 (17.8)
Corneal Fluorescein Staining (CFS) [Mean (Standard Deviation); unit: units on a scale] — The Corneal Fluorescein Staining (CFS) scale ranges from 0 to 15 scale, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of epitheliopathy.
  units on a scale | 1.9 (1.6) | 2.0 (2.0) | 0.9 (1.0) | 1.6 (1.6)
Tear Film Break-Up Time (TBUT) [Mean (Standard Deviation); unit: Seconds] — TBUT measures the amount of time, in seconds, a dry spot appears in the tear film after each blink. Values less than 10 seconds are considered abnormal.
  Seconds | 2.9 (1.5) | 3.0 (1.5) | 2.3 (2.5) | 3.0 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index (OSDI)
Description: A 12-question survey used to measure the symptoms of dry eye disease. Each of the 12 individual questions rate one symptom on a 0-4 scale, with 4 meaning that the symptom is present all of the time and 0 meaning the symptom is present none of the time. The overall ODSI score is calculated by adding all of the values from the 12 questions, multiplying that value by 25, and dividing the resulting value by the number of questions answered. This results in an overall scale that ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms.
Time Frame: 4 week Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide
Number analyzed (Participants) | 13 | 14 | 14
units on a scale | 38.7 (20.3) | 36.9 (28.2) | 37.3 (21.0)

2. Primary Outcome: Symptom Assessment in Dry Eye (SANDE)
Description: A two-item survey used to assess the frequency and severity of dry eye disease. The SANDE score is calculated by taking the square root of the product of the frequency of symptoms score and the severity of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: 4 week Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide
Number analyzed (Participants) | 13 | 14 | 14
units on a scale | 49.1 (22.5) | 50.2 (27.6) | 47.6 (25.5)

3. Primary Outcome: Corneal Fluorescein Staining (CFS)
Description: Is used to assess the level of corneal epitheliopathy that is related to dry eye disease. The CFS scale ranges from 0 to 15 scale, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of epitheliopathy.
Time Frame: 4 week Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide
Number analyzed (Participants) | 13 | 14 | 14
units on a scale | 2.4 (2.4) | 2.0 (2.2) | 1.4 (2.1)

4. Primary Outcome: Tear Break Up Time (TBUT)
Description: TBUT measures the amount of time, in seconds, a dry spot appears in the tear film after each blink. Values less than 10 seconds are considered abnormal.
Time Frame: 4 week Time Point
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide
Number analyzed (Participants) | 13 | 14 | 14
Seconds | 3.5 (2.4) | 4.2 (3.0) | 3.2 (2.9)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Meibomian Gland Probing Plus Lubricant | Sham Meibomian Gland Probing Plus Lubricant | Meibomian Gland Probing Plus Blephamide
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/13 | 3/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Meibomian Gland Probing Plus Lubricant (N=13) | Sham Meibomian Gland Probing Plus Lubricant (N=14) | Meibomian Gland Probing Plus Blephamide (N=14)
Eye Pain (Eye disorders) | 1 | 1 | 2
Redness (Eye disorders) | 0 | 2 | 0
Foreign Body Sensation (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes